CLINICAL TRIAL: NCT03795779
Title: Phase I, Interventional, Single Arm, Open Label, Treatment Study to Evaluate The Safety and Tolerability of CLL1-CD33 cCAR in Patients With Relapsed and/or Refractory, High Risk Hematologic Malignancies.
Brief Title: CLL1-CD33 cCAR in Patients With Relapsed and/or Refractory, High Risk Hematologic Malignancies
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: iCell Gene Therapeutics (Industry)
Collaborators: The General Hospital of Western Theater Command (Other); iCAR Bio Therapeutics Ltd. (Industry); Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICG141-001
Record Dates: First submitted 2019-01-02; First posted 2019-01-08 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Hematologic Malignancy; Acute Myeloid Leukemia; Myelodysplastic Syndromes; Myeloproliferative Neoplasm; Chronic Myeloid Leukemia
Keywords: CLL1; CD33; CLL1-CD33 cCAR; Leukemia; Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLL1-CD33 cCAR T cells (Experimental): CLL1-CD33cCAR T cells transduced with a lentiviral vector to express two distinct units of anti-CLL1 and CD33 CARs
  Interventions: Biological: CLL1-CD33 cCAR T cells

INTERVENTIONS:
Biological: CLL1-CD33 cCAR T cells — CLL1-CD33 cCAR T cells transduced with a lentiviral vector to express two distinct units of anti-CLL1 and CD33 CARs.

SUMMARY:
Phase I, interventional, single arm, open label, treatment study to evaluate the safety and tolerability of CLL1-CD33 cCAR in patients with relapsed and/or refractory, high risk hematologic malignancies.

DETAILED DESCRIPTION:
AML bears heterogeneous cells that can consequently offset killing by single-CAR-based therapy, which results in disease relapse. Leukemic stem cells (LSCs) associated with CLL1 expression comprise a rare population that also plays an important role in disease progression and relapse for myeloid malignancies. CD33 is widely expressed in AML, high risk myelodysplastic syndromes (MDS) and myeloproliferative neoplasms. Targeting both CD33 and CLL1 surface antigens together may offer two distinct benefits. First, targeting both bulk disease and leukemic stem cells together allows for a more comprehensive ablation of the disease. Second, dual targeting of myeloid malignancies by both CD33 and CLL1 directed therapy overcomes the pitfalls of single-antigen therapy by preventing relapse due to antigen loss. While loss of a single antigen under antigen-specific selection pressure is possible, loss of two antigens simultaneously is much less likely.

CLL1-CD33 cCAR is a compound Chimeric Antigen Receptor (cCAR) immunotherapy with two distinct functional CAR molecules expressed on a T-cell, directed against the surface proteins CLL1 and CD33. cCAR intends to target the mechanisms of single-CAR relapse, specifically antigen escape and leukemic stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. Prior HSCT relapse beyond 6 months without active GVHD; systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 4 weeks
2. De novo AML
3. Transformed AML
4. MDS with excess blasts (RAEB-2)
5. MDS that is not a candidate for induction chemotherapy.
6. Myeloproliferative neoplasms with blastic transformation
7. Patients have exhausted standard therapeutic options

Exclusion Criteria:

1. Prior solid organ transplantation
2. Potentially curative therapy including hematopoietic cell transplant
3. Prior treatment with CD123xCD3 or CLL1x3 bispecific agents, T cells expressing CD123 CAR or CLL1 CAR, or toxin-conjugated to CD123 or CLL1 antibodies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicity (DLT) as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 28 days
Type of dose-limiting toxicity (DLT) | 28 days
Number of participants with adverse event by severity as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 2 years

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  Assessment of morphologic complete remission (CR), complete remission with incomplete recovery of counts (CR1), no residual disease as analyzed by flow cytometry analysis, and molecular remission by molecular studies
Progression-free survival (PFS) | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Zhang, MD, PhD, Principal Investigator — Peking University Shenzhen Hospital; Fang Liu, MD, PhD, Principal Investigator — The General Hospital of Western Theater Command
Locations (2):
- China (2):
  - The General Hospital of Western Theater Command, Chengdu
  - Peking University Shenzhen Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No